CLINICAL TRIAL: NCT04005508
Title: Prospective Study on Obstructive Sleep Apnea and Cardiovascular Outcomes in Patients With Atrial Fibrillation and High Cardiovascular Risk
Brief Title: OSA and CV Outcomes in Patients With High Risk AF
Acronym: POACH
Status: Recruiting | Type: Observational
Sponsor: National University of Singapore (Other)
Collaborators: Ng Teng Fong General Hospital (Other); National University Hospital, Singapore (Other); Singapore General Hospital (Other)
Responsible Party: Principal Investigator, Chi-Hang Lee, Professor, National University of Singapore
Other Study IDs: POACH
Record Dates: First submitted 2019-06-29; First posted 2019-07-02 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Atrial Fibrillation; Obstructive Sleep Apnea
Keywords: sleep; cardiovascular outcomes; high cardiovascular risk; observational
MeSH Terms: conditions — Atrial Fibrillation; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OSA (Watch PAT AHI >/= 15 events per hour): Patients found to have OSA by an overnight sleep study
  Interventions: Diagnostic Test: Overnight sleep study
- Non-OSA (Watch PAT AHI < 15 events per hour): Patients found NOT to have OSA by an overnight sleep study
  Interventions: Diagnostic Test: Overnight sleep study

INTERVENTIONS:
Diagnostic Test: Overnight sleep study — The patients will undergo an overnight sleep study using Watch-PAT sleep study device

SUMMARY:
The POACH study is part of the Cardiosleep research program. It is a prospective, observational, multicentre study conducted in Singapore. The recruitment target is 1365 patients.

Eligible patients with AF and high cardiovascular risk will be recruited for a home-based sleep study using a FDA-approved portable device. The patients will be divided into 2 groups based on the presence or absence of OSA using apnoea-hypopnoea index ≥ 15 events/hour. The AF will be treated as per local standard practice. Participation in the POACH study will not affect the management of AF. Follow-up will be conducted every 6 months until the median follow-up duration has reached 2 years. The primary endpoint is a four-component composite of all-cause mortality, myocardial infarction, stroke and heart failure hospitalisation.

Antecubital venous blood samples will be taken from the patients in the morning after the sleep study for targeted mass spectrometry which will measure 83 circulating metabolites. Sparse Principal Component Analysis will be used for data reduction. Identification of distinct associations between metabolic perturbations and OSA will be performed.

DETAILED DESCRIPTION:
The overarching objective of the POACH study is to determine the impact of obstructive sleep apnoea (OSA) on cardiovascular outcomes in patients with atrial fibrillation (AF).

AF is the most prevalent sustained arrhythmia. While OSA often co-exists with AF, current management of AF does not take OSA status into consideration. This is partly due to the lack of data on whether OSA is independently associated with cardiovascular events in patients with AF. Besides, metabolomics is an emerging field of 'omics' research focusing on profiling and quantifying low-molecular weight components.

The POACH study is part of the Cardiosleep research program. It is a prospective, observational, multicentre study conducted in Singapore. The recruitment target is 1365 patients.

Eligible patients with AF and high cardiovascular risk will be recruited for a home-based sleep study using a FDA-approved portable device. The patients will be divided into 2 groups based on the presence or absence of OSA using apnoea-hypopnoea index ≥ 15 events/hour. The AF will be treated as per local standard practice. Follow-up will be conducted every 6 months until the median follow-up duration has reached 2 years. The primary endpoint is a four-component composite of all-cause mortality, myocardial infarction, stroke and heart failure hospitalisation. Antecubital venous blood samples will be taken from the patients in the morning after the sleep study for targeted mass spectrometry which will measure 83 circulating metabolites. Sparse Principal Component Analysis will be used for data reduction. Identification of distinct associations between metabolic perturbations and OSA will be performed.

Results of the POACH study will likely impact the care of patients with AF.

ELIGIBILITY:
Inclusion Criteria:

1. Age 22 or above
2. Known AF, including paroxysmal, persistent or permanent AF
3. High cardiovascular risk, defined as one or more of the following:

   * hypertension
   * diabetes mellitus
   * stroke
   * significant coronary artery disease (at least one stenosis of >50% diameter in at least one major epicardial artery based on CT or conventional coronary angiography, positive stress test [treadmill, myocardial perfusion scan, or stress echocardiography], previous percutaneous coronary intervention, or previous coronary artery bypass surgery)
   * chronic kidney disease (excluding polycystic kidney disease) with an estimated glomerular filtration rate of <60 ml/min/1.73m2,
   * 10-year risk of cardiovascular disease of 15% or greater on the basis of the Framingham risk score, or
   * age of 75 years or older

Exclusion Criteria:

1. Known OSA on regular CPAP treatment
2. Valvular AF (moderate/severe mitral stenosis or mechanical heart valve)
3. Permanent pacemaker implantation
4. Life expectancy less than 1 year based on concomitant medical conditions
5. Unable to give research consent
6. Pregnant or lactating women

Ages: 22 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AF and high cardiovascular risk
Sampling Method: Non-Probability Sample
Enrollment: 1365 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | 5 years
  Composite of all-cause mortality, myocardial infarction, stroke and heart failure hospitalization

SECONDARY OUTCOMES:
All-cause mortality | 5 years
  Death due to any cause
All-cause mortality, myocardial infarction, or stroke | 5 years
  tripe composite endpoint
Cardiovascular death | 5 years
  Death due to cardiovascular cause
Cardiovascular death, myocardial infarction, or stroke | 5 years
  tripe composite endpoint
Ischemic stroke | 5 years
  Stroke is defined as global or focal cerebral, spinal cord or retinal injury resulting in acute neurological dysfunction due to ischemia
Heart failure hospitalisation | 5 years
  the presence of congestive heart failure being the primary disease process accounting for clinical and physical signs of heart failure, with a need for additional or increased heart failure therapy, requiring at least a 24 hour stay in an inpatient unit or emergency department
Recurrence of AF after attempts at rhythm control | 5 years
  Recurrence of AF after attempts at rhythm control (pharmacological, catheter, or cardioversion)
AF Progression | 5 years
  Defined as (1) paroxysmal AF at baseline becoming persistent or permanent at the last follow-up visit or (2) persistent AF at baseline becoming permanent at the last follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Hang R Lee, MD, Principal Investigator — National University of Singapore
Locations (1):
- Chi-Hang Lee, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No